CLINICAL TRIAL: NCT05406440
Title: A Multiple Ascending Dose Clinical Study to Evaluate the Safety, Tolerability, PK and the Effect of MK-8189 on QTc in Participants With Schizophrenia
Brief Title: A Study of MK-8189 in Participants With Schizophrenia (MK-8189-014)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8189-014; MK-8189-014 (Other: Merck)
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Results first posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — MK-8189

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MK-8189 Panel A (Experimental): Participants will receive MK-8189 starting at 48 mg on Day 1 and 60 mg on Day 2.
  Interventions: Drug: MK-8189
- MK-8189 Panel A-1 (Experimental): Participants will receive MK-8189 48 mg on Day 1 and 80 mg on Day 2.
  Interventions: Drug: MK-8189
- MK-8189 Panel C (Experimental): Participants will receive MK-8189 48 mg on Days 1-2 and 80 mg on Day 3 based on safety and tolerability.
  Interventions: Drug: MK-8189
- Placebo (Placebo Comparator): Participants will receive MK-8189-matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-8189 — MK-8189 4 mg and/or 12 mg tablet(s) will be administered orally QD for a total daily dose of 48 mg, 60 mg, 80 mg.
  Arms: MK-8189 Panel A; MK-8189 Panel A-1; MK-8189 Panel C
Drug: Placebo — MK-8189 dose-matching placebo tablets will be administered orally QD.
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to assess the safety and tolerability of multiple ascending doses of MK-8189 in participants with schizophrenia.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Meets diagnostic criteria for schizophrenia or schizoaffective disorder according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria with the onset of the first episode being no less than 2 years prior to screening and monotherapy with antipsychotics for treatment should be indicated.
* Is in the non-acute phase of their illness and clinically stable for 3 months prior to screening as demonstrated by: 1) no clinically significant change in dose of prescribed antipsychotic medication, or clinically significant change in antipsychotic medication to treat symptoms of schizophrenia for two months prior to screening; 2) no increase in level of psychiatric care due to worsening of symptoms of schizophrenia for three months prior to screening.
* Has a history of receiving and tolerating antipsychotic medication within the usual dose range employed for schizophrenia.
* Is able to discontinue the use of all antipsychotic medication at least 5 days or 3 half-lives (whichever is longer) prior to Day -1 and during the study period.

Exclusion Criteria:

* Is at imminent risk of self-harm.
* Has a history of cancer (malignancy). Exceptions: 1) adequately treated nonmelanomatous skin carcinoma or carcinoma in situ of the cervix; 2) malignancies which have been successfully treated ≥10 years prior to the prestudy (screening) visit; 3) highly unlikely to sustain a recurrence for the duration of the study.
* Has evidence or history of a primary DSM-5 axis I psychiatric diagnosis other than schizophrenia or schizoaffective disorder per the allowed DSM-5 criteria within one month of screening.
* Has evidence or history of mental retardation, borderline personality disorder, anxiety disorder, or organic brain syndrome.
* Has a history of neuroleptic malignant syndrome or moderate to severe tardive dyskinesia.
* Has a substance-induced psychotic disorder or behavioral disturbance thought to be due to substance abuse.
* Has a DSM-5 defined substance use disorder (excluding nicotine and caffeine) within 3 months of screening.
* Has a history of seizure disorder beyond childhood or is receiving treatment with any anticonvulsant to prevent seizures.
* Has a clinically significant history or presence of sick sinus syndrome, first, second, or third degree atrioventricular (AV) block, myocardial infarction, pulmonary congestion, cardiac arrhythmia, prolonged corrected QT (QTc) interval, or conduction abnormalities.
* Meets any of the following cardiac parameters: a history of risk factors for Torsades de Pointes (eg, heart failure/cardiomyopathy or family history of long QT syndrome), uncorrected hypokalemia or hypomagnesemia, or is taking concomitant medications that prolong the QT/QTc interval.
* Has history of repeated or frequent syncope, vasovagal episodes, or epileptic seizures.
* Has a family history of cardiac sudden death.
* Is positive for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus (HIV).
* Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the prestudy (screening) visit.
* Has received or is currently receiving treatment with clozapine for schizophrenia for any length of time or treatment with monoamine oxidase inhibitors within 3 months of screening or cariprazine within 2 months of screening.
* Has received a parenteral depot antipsychotic medication within 3 months of screening.
* Has received any nonlive vaccine starting from 14 days prior to study intervention or is scheduled to receive any nonlive vaccine through 30 days following study intervention.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (3):
- United States (3):
  - Collaborative Neuroscience Research, LLC ( Site 0004), Garden Grove, California
  - California Clinical Trials Medical Group managed by PAREXEL ( Site 0002), Glendale, California
  - Hassman Research Institute Marlton Site ( Site 0003), Marlton, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Fifty-three schizophrenia participants randomized to either MK-8189 or placebo in Panels A, A-1, and C. MK-8189 dose and schedule were modified for participants based on saftey and tolerability.
Groups:
- Panel A MK-8189 48-60 mg: Participants with Schizophrenia received monotherapy MK-8189 oral dose of 48 mg QD starting on Day 1 and 60 mg QD on Day 2.
- Panel A Placebo; Panel A-1 Placebo: Participants with Schizophrenia received MK-8189-matching placebo oral dose of 0 mg QD on Day 1 and Day 2.
- Panel A-1 MK-8189 48-80 mg: Participants with Schizophrenia received monotherapy MK-8189 oral dose of 48 mg QD starting on Day 1 and 80 mg QD on Day 2.
- Panel C MK-8189 48-80 mg: Participants with Schizophrenia received monotherapy MK-8189 oral dose of 48 mg QD on Days 1-2 and 80 mg QD on Day 3 based on participant safety and tolerability.
- Panel C MK-8189 48 mg: Participants with Schizophrenia received monotherapy MK-8189 oral dose of 48 mg QD on Days 1-2.
- Panel C Placebo: Participants with Schizophrenia received MK-8189-matching placebo oral dose of 0 mg QD Days 1-3.
Period: Overall Study
Arm/Group | Panel A MK-8189 48-60 mg | Panel A Placebo | Panel A-1 MK-8189 48-80 mg | Panel A-1 Placebo | Panel C MK-8189 48-80 mg | Panel C MK-8189 48 mg | Panel C Placebo
Started | 8 | 3 | 8 | 2 | 18 | 2 | 12
Completed | 8 | 3 | 8 | 2 | 15 | 0 | 12
Not Completed | 0 | 0 | 0 | 0 | 3 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panel A MK-8189 48-60 mg | Panel A Placebo | Panel A-1 MK-8189 48-80 mg | Panel A-1 Placebo | Panel C MK-8189 48-80 mg | Panel C MK-8189 48 mg | Panel C Placebo | Total
Number analyzed (Participants) | 8 | 3 | 8 | 2 | 18 | 2 | 12 | 53
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.1 (9.2) | 42.0 (4.0) | 47.5 (9.7) | 36.0 (4.2) | 42.4 (8.1) | 47.0 (0.0) | 46.1 (8.1) | 44.6 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 4 | 0 | 5 | 2 | 4 | 20
  Male | 4 | 2 | 4 | 2 | 13 | 0 | 8 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 0 | 2 | 0 | 3 | 8
  Not Hispanic or Latino | 7 | 3 | 6 | 2 | 16 | 2 | 9 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 4
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 3 | 6 | 2 | 12 | 2 | 7 | 39
  White | 0 | 0 | 2 | 0 | 2 | 0 | 3 | 7
  More than one race | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporarily associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experienced one or more AEs were reported.
Time Frame: Up to approximately 17 days
Population: All participants who received as least one dose of the investigational drug. Per protocol, safety was assessed by dose.
Measure: Number; unit: Participants
Groups:
- Panel A MK-8189 48 mg: Participants with Schizophrenia received monotherapy MK-8189 oral dose of 48 mg QD on Day 1.
- Panel A MK-8189 60mg; Panel A-1 MK-8189 80 mg: Participants with Schizophrenia received monotherapy MK-8189 oral dose of 80 mg QD on Day 2.
- Panel A-1 MK-8189 48 mg: Participants with Schizophrenia received monotherapy MK-8189 oral dose of 48 mg QD starting on Day 1.
- Panel C MK-8189 48 mg: Participants with Schizophrenia received monotherapy MK-8189 oral dose of 48 mg QD on Days 1-2 based on participant safety and tolerability.
- Panel C MK-8189 80 mg: Participants with Schizophrenia received monotherapy MK-8189 oral dose of 80 mg QD on Day 3 based on participant safety and tolerability.
Arm/Group | Panel A MK-8189 48 mg | Panel A MK-8189 60mg | Panel A Placebo | Panel A-1 MK-8189 48 mg | Panel A-1 MK-8189 80 mg | Panel A-1 Placebo | Panel C MK-8189 48 mg | Panel C MK-8189 80 mg | Panel C Placebo
Number analyzed (Participants) | 8 | 8 | 3 | 8 | 8 | 2 | 20 | 18 | 12
Participants | 3 | 2 | 0 | 3 | 4 | 0 | 7 | 6 | 6

2. Primary Outcome: Number of Participants Who Discontinue From Study Treatment Due to an AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporarily associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinued study due to an AE were reported.
Time Frame: Up to approximately 3 days
Population: All participants who received as least one dose of the investigational drug. Per protocol, safety was assessed by dose.
Measure: Number; unit: Participants
Groups:
- Panel C MK-8189 48 mg: chizophrenia received monotherapy MK-8189 oral dose of 48 mg QD on Days 1-2 based on participant safety and tolerability.
Arm/Group | Panel A MK-8189 48 mg | Panel A MK-8189 60mg | Panel A Placebo | Panel A-1 MK-8189 48 mg | Panel A-1 MK-8189 80 mg | Panel A-1 Placebo | Panel C MK-8189 48 mg | Panel C MK-8189 80 mg | Panel C Placebo
Number analyzed (Participants) | 8 | 8 | 3 | 8 | 8 | 2 | 20 | 18 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 17 days
Description: All participants who received at least one dose of treatment were included
Groups:
- Panel A MK-8189 Dose 48 mg: Participants with Schizophrenia received monotherapy MK-8189 oral dose of 48 mg QD on Day 1.
Arm/Group | Panel A MK-8189 Dose 48 mg | Panel A MK-8189 60mg | Panel A Placebo | Panel A-1 MK-8189 48 mg | Panel A-1 MK-8189 80 mg | Panel A-1 Placebo | Panel C MK-8189 48 mg | Panel C MK-8189 80 mg | Panel C Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/3 | 0/8 | 0/8 | 0/2 | 0/20 | 0/20 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/3 | 0/8 | 0/8 | 0/2 | 0/20 | 0/18 | 0/12
Other Adverse Events (participants affected / at risk) | 3/8 | 2/8 | 0/3 | 3/8 | 4/8 | 0/2 | 7/20 | 6/18 | 6/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panel A MK-8189 Dose 48 mg (N=8) | Panel A MK-8189 60mg (N=8) | Panel A Placebo (N=3) | Panel A-1 MK-8189 48 mg (N=8) | Panel A-1 MK-8189 80 mg (N=8) | Panel A-1 Placebo (N=2) | Panel C MK-8189 48 mg (N=20) | Panel C MK-8189 80 mg (N=18) | Panel C Placebo (N=12)
Miosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Akathisia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dystonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Nystagmus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oromandibular dystonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Substance use (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT05406440/Prot_SAP_000.pdf